CLINICAL TRIAL: NCT05846269
Title: A Resiliency and Trauma-Informed Care Intervention for Psychiatric Mental Health Nurse Practitioner Specialty Doctor of Nursing Practice Students
Brief Title: A Resiliency and TIC Intervention for PMHNP Specialty DNP Students
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00002213
Record Dates: First submitted 2022-12-12; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Stress; Trauma
Keywords: Graduate nursing students; Resiliency; Trauma informed care
MeSH Terms: conditions — Wounds and Injuries | interventions — Early Intervention, Educational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2023 Clinical Cohort: Students in the Doctor of Nursing Practice (DNP) nurse practitioner specialties and certificate programs in the clinical year of their programs during 2023.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Educational intervention addressing trauma-informed care and resiliency.

SUMMARY:
The goal of this observational study is to explore the impact of a resiliency and trauma informed care educational intervention for Psychiatric Mental Health Nurse Practitioner (PMHNP) students at the University of Arizona College of Nursing during the final, clinical year of the program. Specifically, the investigators will examine if the educational intervention is feasible, acceptable and helpful to students, and can decrease burnout and increase resiliency.

DETAILED DESCRIPTION:
Students in the Doctor of Nursing Practice (DNP) and certificate programs during their final, clinical year of the program will be asked to complete anonymous online surveys before each semester (Spring, Summer, and Fall) that measure levels of burnout, resiliency, Adverse Childhood Experiences (ACEs), perceived stress, and knowledge related to trauma-informed care principles and ways to promote their resiliency. Students in the Psychiatric Mental Health Nurse Practitioner (PMHNP) specialty will receive an educational intervention related to trauma-informed care and resiliency during an in-person clinical immersion in January, May, and August 2023; after each session, they will be asked to complete an anonymous online post-intervention survey. Each survey includes a disclosure statement and list of University and national mental health resources in case participants experience any emotional distress related to the topics/questions related to the survey.

ELIGIBILITY:
Inclusion Criteria:

* Doctor of Nursing Practice (DNP) and post-Masters certificate students at the University of Arizona College of Nursing in the final, clinical year of their program.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inclusion criteria will be Doctor of Nursing Practice and Post-Masters certificate students at the University of Arizona College of Nursing. All study participants will be over age 18. The investigators will include participants of all genders and ethnicities that meet our inclusion criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Trauma informed care knowledge questionnaire | 2023 Academic Year
  An original online survey designed by the investigators to align with objectives of intervention and to measure participants' knowledge and confidence related to trauma informed care principles. Composed of 12 items, all open-ended or Likert scale responses.
Resiliency knowledge and skills questionnaire | 2023 Academic Year
  An original online survey designed by the investigators to align with objectives of intervention and to measure participants' knowledge and confidence related to trauma informed care principles. Composed of 12 items, all open-ended or Likert scale responses.

SECONDARY OUTCOMES:
Maslach Burnout Inventory Scale questionnaire | 2023 Academic Year
  Min value=0, max value=132, higher score indicates more professional burnout (worse outcome)
Connor-Davison Resilience Scale 25 (CD-RISC-25) questionnaire | 2023 Academic Year
  Min value=0, max value=100, higher score indicates better resiliency (better outcome)
Perceived Stress Scale questionnaire | 2023 Academic Year
  Min value=0, max value=40, higher score indicates higher perceived stress (worse outcome)
Adverse Childhood Experiences (ACEs) questionnaire | Spring 2023
  Min value=0, max value=10, higher score indicates more negative childhood experiences related to physical and mental health issues later in life (worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Bouchard, DNP, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No